CLINICAL TRIAL: NCT05196191
Title: Randomized Control Trial of Vivex Tissue for Accelerated Wound Healing Following Penile Prosthesis Placement With Follow-up
Brief Title: Wound Healing Following Penile Prosthesis Implant
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: VIVEX Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CYG-2021-001
Record Dates: First submitted 2021-12-14; First posted 2022-01-19 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Erectile Dysfunction
Keywords: Viagenex Max; penile implant; erectile dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: Subjects meeting criteria will be randomized 4:1 treatment (Viagenex Max) or sham (standard of care).
Who Masked: Participant
Masking Description: Subjects will not be told which treatment group they receive until the end of study participation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Viagenex Max (Experimental): VIAGENEX Max graft will be placed in the incision at the end of surgery prior to closing.
  Interventions: Biological: VIAGENEX Max
- Standard of care (Active Comparator): Hibiclens wash will be performed.
  Interventions: Procedure: Hibiclens wash

INTERVENTIONS:
Biological: VIAGENEX Max — Collagenous membrane derived from umbilical cord
  Arms: Viagenex Max
Procedure: Hibiclens wash — Antiseptic skin cleanser
  Arms: Standard of care

SUMMARY:
This is a prospective, randomized, clinical study aimed to evaluate the safety and efficacy of the two treatment schedules on men undergoing penile implant surgery for the first time. The patients are randomized in a 2:1 ratio of active to sham treatment groups.

DETAILED DESCRIPTION:
Erectile Dysfunction (ED) is a condition with an inability to develop or maintain an erection of the penis upon sexual stimulation. It occurs in association with aging, chronic illnesses and various modifiable risk factors. Amongst the modifiable risk factors, ED shares the most common risk factors with Coronary Artery Disease (CAD) which are smoking, hypertension and hyperlipidemia. Even though it is not a part of normal aging, it is seen in 52% of men in the age group 40 to 70 years, with a higher rate in the men more than 70 years.

VIAGENEX Max is a semi-transparent, collagenous membrane intended for soft tissue barrier or wound covering, derived from umbilical cord membrane. A total of 50 subjects with ED meeting the eligibility criteria will be randomized. The treatment graft will be placed into the wound at time of surgery. The treatment group will receive the VIAGENEX graft and the sham group will receive the standard of care for this surgery.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be willing and able to provide informed consent
* The patient is a male between >/= 30 and =/< 70 years of age
* The patient has ED based of International Index of Erectile Dysfunction (IIEF) scores
* The patient has been in a stable relationship for over 3 months prior to enrollment
* A minimum of 2 sexual attempts per month for at least one month prior to enrollment - as documented by IIEF
* The patient is suffering from erectile dysfunction and undergoing penile implant surgery for the first time
* IIEF-EF score between 16 and 25
* Testosterone level 300-1000 ng/dL within 1 month prior to enrollment
* A1C level </= 7% within 1 month prior to enrollment

Exclusion Criteria:

* The patient is currently or has participated in another study within the past three months that may interfere with the results or conclusions of this study
* The patient is under judicial protection (prison or custody)
* The patient is an adult under guardianship
* The patient refuses to sign the consent
* History of radical prostatectomy or extensive pelvic surgery
* Evidence of venous leak
* Past radiation therapy of the pelvic region within 12 months prior to enrollment
* Recovering from any cancer within 12 months prior to enrollment
* Neurological disease such as Alzheimer's or Parkinson's disease which affects erectile function at the discretion of the investigator
* Psychiatric diagnosis or medications such as antidepressants, anxiolytic, antipsychotic that affects erectile function or any other medications at the discretion of the investigator
* Anatomical malformation of the penis, including Peyronie's disease
* Testosterone level <300 or >1000 ng/dL within 1 month prior to enrollment
* A1C level > 7% within 1 month prior to enrollment or history of insulin dependent diabetes
* The patient is taking blood thinners and has an international normalized ratio >3
* Received shockwave treatment at least 6 months before enrollment

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 32 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Penile implant activation | up to 3 months
  Time to use implant for sexual activity

SECONDARY OUTCOMES:
Pain after undergoing penile prosthesis surgery | surgery to 12 months
  Numerical pain scale (0=no pain to 10=worst pain) used to

CONTACTS AND LOCATIONS:
Overall Officials: Tariq Hakky, MD, Principal Investigator — Atlanta Cosmetic Urology
Locations (1):
- Atlanta Cosmetic Urology, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.